CLINICAL TRIAL: NCT03229538
Title: STeroids to REduce Systemic Inflammation After Infant Heart Surgery (STRESS)
Brief Title: STeroids to REduce Systemic Inflammation After Infant Heart Surgery
Acronym: STRESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kevin Hill (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Kevin Hill, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00078106; 1U01TR001803-01 (NIH)
Record Dates: First submitted 2017-07-05; First posted 2017-07-25 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2023-05

CONDITIONS: Congenital Heart Disease in Children; Inflammatory Response
MeSH Terms: interventions — Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone Arm (Experimental): IV Methylprednisolone
  Interventions: Drug: Methylprednisolone
- Placebo Arm (Placebo Comparator): IV Isotonic Saline
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Methylprednisolone — IV Steroid pre-operative and intra-operative
  Arms: Methylprednisolone Arm
Drug: Isotonic saline — Isotonic saline pre-operative and intra-operative
  Arms: Placebo Arm

SUMMARY:
This study's objective is to determine the pharmacokinetics (PK)/pharmacodynamics (PD), safety and efficacy of methylprednisolone in infants undergoing heart surgery with cardiopulmonary bypass. This is a prospective, double blind, multi-center, placebo-controlled safety and efficacy study. Blood samples will be collected from a subset of enrolled study participants to evaluate multiple dose methylprednisolone PK/PD. Participants will be randomized in a 1:1 fashion to intravenous methylprednisolone versus placebo. Study drug/placebo will be administered 8 to 12 hours before the anticipated start time of surgery and in the operating room at the time of initiation of cardiopulmonary bypass. Patients will be followed for primary and secondary outcomes for the duration of their hospitalization. Serious study drug-related adverse events will be collected for 7 days after the last dose of study drug.

DETAILED DESCRIPTION:
Overview:

Congenital heart diseases (CHD) are the most common birth defects, occurring in nearly 1% of live births. Every year, an estimated 40,000 infants born in the U.S. suffer from CHD. Despite advances in surgical management, CHD requiring neonatal surgery is associated with poor outcomes; national registry data demonstrates post-operative major morbidity in 23% and 10% do not survive to hospital discharge.

Poor outcomes after neonatal heart surgery are often attributable to a severe systemic inflammatory response to cardiopulmonary bypass (CPB). CPB is necessary for most neonatal CHD surgeries. Therefore, to reduce the post-CPB inflammatory reaction, many surgeons administer pre-or intra-operative steroids. Steroids have been shown to reduce inflammatory markers after neonatal heart surgery. However, steroids also have potential harmful effects including an increased risk of post-operative infection. The recent SIRS trial evaluated the safety and efficacy of steroids after CPB in adults and demonstrated no beneficial effect of steroids but increased risk of post-CPB myocardial infarction and other major adverse events.

Adult trial results cannot be reliably extrapolated to neonates because the neonatal response to CPB is markedly different to that seen in adults; neonates demonstrate both a more pronounced inflammatory reaction and a different post-operative complication profile. For these reasons approximately 2/3rds of congenital heart surgeons continue to administer perioperative steroids to neonates undergoing heart surgery. Yet this practice is not evidence based as no safety/efficacy trial has ever evaluated steroids in neonates undergoing heart surgery with CPB. Several smaller steroid trials (all enrolling < 75 patients) have focused on surrogate outcome measures, but none have provided conclusive data.

The major barrier to performing a steroid trial in neonates with CHD has been the high cost associated with trial conduct for these relatively rare defects. To overcome this barrier, the investigators will use a novel approach leveraging existing registry infrastructure at CHD surgical sites that participate in the Society of Thoracic Surgeons Congenital Heart Surgery Database (STS-CHSD). Sites participating in the STS-CHSD collect data into their institutional databases using standardized case report forms so that the data can be exported to the STS-CHSD. These sites already employ data coordinating specialists to capture patient demographics, procedural variables, and post-operative outcomes (including a list of over 60 complication variables) using strict and consistent data element definitions. By leveraging these site-specific resources the investigators project that the investigators can reduce trial costs by >75%.

Background:

Some surgeons/centers currently administer perioperative high dose (20mg to 60mg) intravenous methylprednisolone before neonatal heart surgery with CPB. In a national registry study of > 3000 neonates with data capture spanning 2004 to 2008, 62% of neonates undergoing surgery with CPB received perioperative methylprednisolone while 38% did not. Of those receiving methylprednisolone, 22% received methylprednisolone on both the day before, and day of surgery, 12% on the day before surgery only, and 28% on the day of surgery only. Results of a survey of surgeons from the Congenital Heart Surgeon's Society were similar; 28% did not routinely use steroids for neonatal heart surgery. Of the 72% that did routinely use steroids, ~1/3rd administered steroids pre-operatively and intra-operatively and the remainder gave intra-operative steroids only.

Several previous small translationally focused clinical trials have evaluated the safety and efficacy of methylprednisolone. In the largest contemporary trial, neonates scheduled for cardiac surgery were prospectively randomized to receive either 2-dose (8 hours preoperatively and operatively, n = 39) or single-dose (operatively, n = 37) methylprednisolone at 30 mg/kg IV per dose in a prospective double-blind trial. Neonates receiving pre-operative methylprednisolone therapy demonstrated significantly reduced pre-operative pro-inflammatory cytokines including interleukin-6 and 8. There were no differences between the two groups in post-operative pro-inflammatory markers and no differences in the incidence of post-operative low cardiac output syndrome. Methylprednisolone was well tolerated with no adverse drug reactions. The overall incidence of post-operative infection was 13% (10/76) and 4% (3/76) received a post-operative insulin infusion for hyperglycemia.

A meta-analysis evaluated six previous steroid trials in children undergoing heart surgery with CPB. The combined enrollment of these six trials was 232 participants including 116 receiving peri-operative steroids; two of these studies used methylprednisolone at doses of 30mg/kg IV per dose (n=67 patients). The results of this meta-analysis demonstrated a nonsignificant trend of reduced mortality in steroid-treated patients (11 [4.7%] vs 4 [1.7%] patients; odds ratio, 0.41; 95% CI, 0.14-1.15; p = 0.089). Steroids had no effects on mechanical ventilation time (117.4 ± 95.9 hr vs 137.3 ± 102.4 hr; p = 0.43) and ICU length of stay (9.6 ± 4.6 d vs 9.9 ± 5.9 d; p = 0.8). Perioperative steroid administration reduced the prevalence of renal dysfunction (13 [54.2%] vs 2 [8%] patients; odds ratio, 0.07; 95% CI, 0.01-0.38; p = 0.002). There were no significant differences in the adverse event profiles for patients receiving steroids versus placebo.

The conclusions of the aforementioned studies, as well as several associated editorials have all been that a large, randomized, controlled trial is needed to evaluate the safety and efficacy of perioperative steroids for neonatal heart surgery with CPB.

Design:

This study is a prospective, double-blind, multi-center, placebo-controlled safety and efficacy study of methylprednisolone in neonates undergoing heart surgery with CPB. The study will enroll up to 1500 neonates (< 30 days of age) and the total study duration is expected to be approximately 48 months. An ancillary PK/PD/Biomarker study will enroll subjects at select centers. This study is unique in that it is designed to leverage existing registry infrastructure at participating sites so as to reduce trial costs. Participants will be randomized and will receive a randomization ID. This ID will also serve as a unique patient identifier allowing us to crosslink datasets. Participants will then receive two doses of study drug/placebo. The first dose will be administered 8 to 12 hours before anticipated heart surgery and the second dose will be administered into the pump prime during cardiopulmonary bypass. All study participants will then receive routine post-operative care. Participating centers will enter all demographic, preoperative, operative and outcomes data into their existing institutional databases for submission to the STS-CHSD as they currently do. These data will be used to evaluate trial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age < 1 year at the time of surgery
* Undergoing heart surgery with CPB as part of standard clinical care
* Availability and willingness of the parent/legally authorized representative to provide written informed consent

Exclusion Criteria:

* < 37 weeks adjusted gestational age at time of surgery
* Any oral or intravenous steroid treatment within two days of surgery
* Any patient receiving any of the following medications within 2 days of surgery:

Amphotericin B, aminoglutethimide, anticholinesterases, warfarin, P450 3A4 inducers including (but not limited to) carbamazepine, phenobarbital, phenytoin, rifampin, bosentan and nafcillin or P450 3A4 inhibitors including (but not limited to) clarithromycin, voriconazole, itraconazole, ketoconazole, ciprofloxacin, diltiazem, fluconazole, erythromycin and verapamil.

* Infection contraindicating steroid use
* Preoperative mechanical circulatory support or active resuscitation at the time of randomization
* Emergent surgery precluding steroid administration 8-12 hours before surgery

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1263 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hill, Principal Investigator — Duke University
Locations (23):
- United States (23):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Colorado, Denver, Aurora, Colorado
  - University of Florida Health - Shands Hospital, Gainesville, Florida
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Advocate Children's Hospital, Oak Lawn, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital and Medical Center, Omaha, Nebraska
  - Morgan Stanley Children's Hospital of New York Presbyterian, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Texas Children's Hospital, Houston, Texas
  - Utah/Primary Children's Medical Center, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The investigators will disseminate findings through publications, national presentations, participation in the CTSA Consortium, the CTSA website and via the existing infrastructure of the Society of Thoracic Surgeons Congenital Heart Surgery Database. Data collection supported by CTSA funds will follow the principles outlined in the Final NIH Statement on Sharing Research Data. Participating institutions will honor the principle that data sharing is critical for expeditious translation of research findings to the improvement of human health. The investigators abide strictly by the provisions of the Health Insurance Portability and Accountability Act (HIPAA). The investigators will continue to use traditional venues for data sharing, such as publications in leading scientific journals and deposit all applicable NIH-funded research results to PubMed Central in compliance with the NIH's Public Access Policy.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Petrini J, Damus K, Johnston RB Jr. An overview of infant mortality and birth defects in the United States. Teratology. 1997 Jul-Aug;56(1-2):8-10. doi: 10.1002/(SICI)1096-9926(199707/08)56:1/23.0.CO;2-U. No abstract available. PMID 9381406
- [Background] Petrini J, Damus K, Russell R, Poschman K, Davidoff MJ, Mattison D. Contribution of birth defects to infant mortality in the United States. Teratology. 2002;66 Suppl 1:S3-6. doi: 10.1002/tera.90002. PMID 12239736
- [Background] Yang Q, Chen H, Correa A, Devine O, Mathews TJ, Honein MA. Racial differences in infant mortality attributable to birth defects in the United States, 1989-2002. Birth Defects Res A Clin Mol Teratol. 2006 Oct;76(10):706-13. doi: 10.1002/bdra.20308. PMID 17022030
- [Background] Yang Q, Khoury MJ, Mannino D. Trends and patterns of mortality associated with birth defects and genetic diseases in the United States, 1979-1992: an analysis of multiple-cause mortality data. Genet Epidemiol. 1997;14(5):493-505. doi: 10.1002/(SICI)1098-2272(1997)14:53.0.CO;2-2. PMID 9358267
- [Background] Hoffman TM, Wernovsky G, Atz AM, Kulik TJ, Nelson DP, Chang AC, Bailey JM, Akbary A, Kocsis JF, Kaczmarek R, Spray TL, Wessel DL. Efficacy and safety of milrinone in preventing low cardiac output syndrome in infants and children after corrective surgery for congenital heart disease. Circulation. 2003 Feb 25;107(7):996-1002. doi: 10.1161/01.cir.0000051365.81920.28. PMID 12600913
- [Background] Parr GV, Blackstone EH, Kirklin JW. Cardiac performance and mortality early after intracardiac surgery in infants and young children. Circulation. 1975 May;51(5):867-74. doi: 10.1161/01.cir.51.5.867. PMID 235375
- [Background] Wernovsky G, Wypij D, Jonas RA, Mayer JE Jr, Hanley FL, Hickey PR, Walsh AZ, Chang AC, Castaneda AR, Newburger JW, Wessel DL. Postoperative course and hemodynamic profile after the arterial switch operation in neonates and infants. A comparison of low-flow cardiopulmonary bypass and circulatory arrest. Circulation. 1995 Oct 15;92(8):2226-35. doi: 10.1161/01.cir.92.8.2226. PMID 7554206
- [Background] Wan S, LeClerc JL, Vincent JL. Inflammatory response to cardiopulmonary bypass: mechanisms involved and possible therapeutic strategies. Chest. 1997 Sep;112(3):676-92. doi: 10.1378/chest.112.3.676. PMID 9315800
- [Background] Ando M, Park IS, Wada N, Takahashi Y. Steroid supplementation: a legitimate pharmacotherapy after neonatal open heart surgery. Ann Thorac Surg. 2005 Nov;80(5):1672-8; discusison 1678. doi: 10.1016/j.athoracsur.2005.04.035. PMID 16242437
- [Background] Bronicki RA, Backer CL, Baden HP, Mavroudis C, Crawford SE, Green TP. Dexamethasone reduces the inflammatory response to cardiopulmonary bypass in children. Ann Thorac Surg. 2000 May;69(5):1490-5. doi: 10.1016/s0003-4975(00)01082-1. PMID 10881828
- [Background] Checchia PA, Backer CL, Bronicki RA, Baden HP, Crawford SE, Green TP, Mavroudis C. Dexamethasone reduces postoperative troponin levels in children undergoing cardiopulmonary bypass. Crit Care Med. 2003 Jun;31(6):1742-5. doi: 10.1097/01.CCM.0000063443.32874.60. PMID 12794414
- [Background] Clarizia NA, Manlhiot C, Schwartz SM, Sivarajan VB, Maratta R, Holtby HM, Gruenwald CE, Caldarone CA, Van Arsdell GS, McCrindle BW. Improved outcomes associated with intraoperative steroid use in high-risk pediatric cardiac surgery. Ann Thorac Surg. 2011 Apr;91(4):1222-7. doi: 10.1016/j.athoracsur.2010.11.005. PMID 21440149
- [Background] Graham EM, Atz AM, Butts RJ, Baker NL, Zyblewski SC, Deardorff RL, DeSantis SM, Reeves ST, Bradley SM, Spinale FG. Standardized preoperative corticosteroid treatment in neonates undergoing cardiac surgery: results from a randomized trial. J Thorac Cardiovasc Surg. 2011 Dec;142(6):1523-9. doi: 10.1016/j.jtcvs.2011.04.019. Epub 2011 May 20. PMID 21600592
- [Background] Graham EM, Atz AM, McHugh KE, Butts RJ, Baker NL, Stroud RE, Reeves ST, Bradley SM, McGowan FX Jr, Spinale FG. Preoperative steroid treatment does not improve markers of inflammation after cardiac surgery in neonates: results from a randomized trial. J Thorac Cardiovasc Surg. 2014 Mar;147(3):902-8. doi: 10.1016/j.jtcvs.2013.06.010. Epub 2013 Jul 16. PMID 23870160
- [Background] Toledo-Pereyra LH, Lin CY, Kundler H, Replogle RL. Steroids in heart surgery: a clinical double-blind and randomized study. Am Surg. 1980 Mar;46(3):155-60. PMID 7377659
- [Background] Graham EM. The utility of steroids in pediatric cardiac operations*. Pediatr Crit Care Med. 2014 Jun;15(5):492-3. doi: 10.1097/PCC.0000000000000139. No abstract available. PMID 24892482
- [Background] Pasquali SK, Li JS, He X, Jacobs ML, O'Brien SM, Hall M, Jaquiss RD, Welke KF, Peterson ED, Shah SS, Gaynor JW, Jacobs JP. Perioperative methylprednisolone and outcome in neonates undergoing heart surgery. Pediatrics. 2012 Feb;129(2):e385-91. doi: 10.1542/peds.2011-2034. Epub 2012 Jan 23. PMID 22271697
- [Background] Garg AX, Vincent J, Cuerden M, Parikh C, Devereaux PJ, Teoh K, Yusuf S, Hildebrand A, Lamy A, Zuo Y, Sessler DI, Shah P, Abbasi SH, Quantz M, Yared JP, Noiseux N, Tagarakis G, Rochon A, Pogue J, Walsh M, Chan MT, Lamontagne F, Salehiomran A, Whitlock R; SIRS Investigators. Steroids In caRdiac Surgery (SIRS) trial: acute kidney injury substudy protocol of an international randomised controlled trial. BMJ Open. 2014 Mar 5;4(3):e004842. doi: 10.1136/bmjopen-2014-004842. PMID 24598306
- [Background] Scrascia G, Rotunno C, Guida P, Amorese L, Polieri D, Codazzi D, Paparella D. Perioperative steroids administration in pediatric cardiac surgery: a meta-analysis of randomized controlled trials*. Pediatr Crit Care Med. 2014 Jun;15(5):435-42. doi: 10.1097/PCC.0000000000000128. PMID 24717907
- [Background] Jacobs ML, O'Brien SM, Jacobs JP, Mavroudis C, Lacour-Gayet F, Pasquali SK, Welke K, Pizarro C, Tsai F, Clarke DR. An empirically based tool for analyzing morbidity associated with operations for congenital heart disease. J Thorac Cardiovasc Surg. 2013 Apr;145(4):1046-1057.e1. doi: 10.1016/j.jtcvs.2012.06.029. Epub 2012 Jul 24. PMID 22835225
- [Background] Ungerleider RM. Practice patterns in neonatal cardiopulmonary bypass. ASAIO J. 2005 Nov-Dec;51(6):813-5. doi: 10.1097/01.mat.0000183473.93237.10. No abstract available. PMID 16340373
- [Derived] Hill KD, Koerner J, Hong H, Li JS, Hornik C, Kannankeril PJ, Jacobs JP, Baldwin HS, Jacobs ML, Graham EM, Blasiole B, Vener DF, Husain AS, Kumar SR, Benscoter A, Wald E, Karamlou T, Van Bergen AH, Overman D, Eghtesady P, Butts R, Kim JS, Scott JP, Anderson BR, Swartz MF, O'Brien SM. A Bayesian re-analysis of the STRESS trial. Am Heart J. 2026 Feb;292:107282. doi: 10.1016/j.ahj.2025.09.014. Epub 2025 Sep 25. PMID 41015071
- [Derived] Hill KD, Kannankeril PJ, Jacobs JP, Baldwin HS, Jacobs ML, O'Brien SM, Bichel DP, Graham EM, Blasiole B, Resheidat A, Husain AS, Kumar SR, Kirchner JL, Gallup DS, Turek JW, Bleiweis M, Mettler B, Benscoter A, Wald E, Karamlou T, Van Bergen AH, Overman D, Eghtesady P, Butts R, Kim JS, Scott JP, Anderson BR, Swartz MF, McConnell PI, Vener DF, Li JS; STRESS Network Investigators. Methylprednisolone for Heart Surgery in Infants - A Randomized, Controlled Trial. N Engl J Med. 2022 Dec 8;387(23):2138-2149. doi: 10.1056/NEJMoa2212667. Epub 2022 Nov 6. PMID 36342116
- [Derived] Gibbison B, Villalobos Lizardi JC, Aviles Martinez KI, Fudulu DP, Medina Andrade MA, Perez-Gaxiola G, Schadenberg AW, Stoica SC, Lightman SL, Angelini GD, Reeves BC. Prophylactic corticosteroids for paediatric heart surgery with cardiopulmonary bypass. Cochrane Database Syst Rev. 2020 Oct 12;10(10):CD013101. doi: 10.1002/14651858.CD013101.pub2. PMID 33045104
- [Derived] Hill KD, Baldwin HS, Bichel DP, Butts RJ, Chamberlain RC, Ellis AM, Graham EM, Hickerson J, Hornik CP, Jacobs JP, Jacobs ML, Jaquiss RD, Kannankeril PJ, O'Brien SM, Torok R, Turek JW, Li JS; STRESS Network Investigators. Rationale and design of the STeroids to REduce Systemic inflammation after infant heart Surgery (STRESS) trial. Am Heart J. 2020 Feb;220:192-202. doi: 10.1016/j.ahj.2019.11.016. Epub 2019 Dec 9. PMID 31855716
- See also: United States Food and Drug Administration: Pediatric Study Plans: Content of and Process for Submitting Initial Pediatric Study Plans and Amended Initial Pediatric Study Plans Guidance for Industry (Draft). — https://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM360507.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1263 patients consented and randomized; 63 did not receive study drug and are excluded from final analysis.
Groups:
- Methylprednisolone Arm: IV Methylprednisolone
  Methylprednisolone: IV Steroid pre-operative and intra-operative
  Study drug will be administered 8 to 12 hours before the anticipated start time of surgery and in the operating room at the time of initiation of cardiopulmonary bypass.
- Placebo Arm: IV Isotonic Saline
  Isotonic saline: Isotonic saline pre-operative and intra-operative
  Placebo will be administered 8 to 12 hours before the anticipated start time of surgery and in the operating room at the time of initiation of cardiopulmonary bypass.
Period: Overall Study
Arm/Group | Methylprednisolone Arm | Placebo Arm
Started | 599 | 601
Completed | 599 | 601
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylprednisolone Arm | Placebo Arm | Total
Number analyzed (Participants) | 599 | 601 | 1200
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 126 [14 to 191] | 124 [14 to 182] | 125 [14 to 187]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 279 | 267 | 546
  Male | 320 | 334 | 654
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 80 | 63 | 143
  Not Hispanic or Latino | 519 | 538 | 1057
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected on 32 participants.
  Participants
    number analyzed (Participants) | 585 | 583 | 1168
    American Indian or Alaska Native | 5 | 4 | 9
    Asian | 15 | 12 | 27
    Native Hawaiian or Other Pacific Islander | 4 | 0 | 4
    Black or African American | 90 | 102 | 192
    White | 428 | 425 | 853
    More than one race | 13 | 15 | 28
    Unknown or Not Reported | 30 | 25 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 599 | 601 | 1200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants at Each Global Rank Endpoint Based Upon Their Most-severe Outcome
Description: A composite mortality, major morbidity and length of stay global rank endpoint with endpoints ranked according to severity. For this endpoint, each randomized patient will be assigned a rank based upon their most-severe outcome. Rank of 91 = Post-operative length of stay > 90 days, 92 = Post-op cardiac arrest, multi-system organ failure, renal failure with temporary dialysis, or prolonged ventilator support, 93 = Reoperation for bleeding, unplanned delayed sternal closure, or post-op unplanned interventional cardiac catheterization, 94 = Post-operative mechanical circulatory support or unplanned cardiac reoperation (exclusive of reoperation for bleeding), 95 = Renal failure with permanent dialysis, neurologic deficit persistent at discharge, or respiratory failure requiring tracheostomy; 96 = Heart transplant (during hospitalization); 97 = Operative mortality. Ranks 1 through 90 correspond to the post-operative length of stay in days.
Time Frame: Until hospital discharge, up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 599 | 601
Participants
  Rank = 97 | 12 | 17
  Rank = 96 | 3 | 7
  Rank = 95 | 4 | 8
  Rank = 94 | 44 | 36
  Rank = 93 | 12 | 30
  Rank = 92 | 24 | 22
  Rank = 91 | 4 | 2
  Rank = 81-90 | 0 | 1
  Rank = 71-80 | 0 | 0
  Rank = 61-70 | 2 | 5
  Rank = 51-60 | 5 | 3
  Rank = 41-50 | 6 | 7
  Rank = 31-40 | 14 | 18
  Rank = 21-30 | 44 | 46
  Rank = 11-20 | 115 | 112
  Rank = 0-10 | 310 | 287
Statistical Analysis 1: Comparison: Methylprednisolone Arm vs Placebo Arm; Test type: Other; p = 0.14, Regression, Logistic; Adjusted Odds Ratio = 0.86, 95% CI 2-sided [0.71 to 1.05]
Statistical Analysis 2: Comparison: Methylprednisolone Arm vs Placebo Arm; Rank = 97; Test type: Other; Percent Difference = -0.8, 95% CI 2-sided [-2.6 to 0.9] — Difference = Methylprednisolone - Placebo
Statistical Analysis 3: Comparison: Methylprednisolone Arm vs Placebo Arm; Rank > or = 96; Test type: Other; Percent Difference = -1.5, 95% CI 2-sided [-3.5 to 0.5] — Difference = Methylprednisolone - Placebo
Statistical Analysis 4: Comparison: Methylprednisolone Arm vs Placebo Arm; Rank > or = 95; Test type: Other; Percent Difference = -2.2, 95% CI 2-sided [-4.4 to 0.1] — Difference = Methylprednisolone - Placebo
Statistical Analysis 5: Comparison: Methylprednisolone Arm vs Placebo Arm; Rank > or = 94; Test type: Other; Percent Difference = -0.8, 95% CI 2-sided [-4.3 to 2.7] — Difference = Methylprednisolone - Placebo
Statistical Analysis 6: Comparison: Methylprednisolone Arm vs Placebo Arm; Rank > or = 93; Test type: Other; Percent Difference = -3.8, 95% CI 2-sided [-7.8 to 0.2] — Difference = Methylprednisolone - Placebo
Statistical Analysis 7: Comparison: Methylprednisolone Arm vs Placebo Arm; Rank > or = 92; Test type: Other; Percent Difference = -3.4, 95% CI 2-sided [-7.8 to 0.9] — Difference = Methylprednisolone - Placebo
Statistical Analysis 8: Comparison: Methylprednisolone Arm vs Placebo Arm; Rank > or = 91; Test type: Other; Percent Difference = -3.1, 95% CI 2-sided [-7.5 to 1.3] — Difference = Methylprednisolone - Placebo

2. Secondary Outcome: Number of Participants With Mortality, Including In-hospital Mortality or Mortality After Hospital Discharge But Within 30 Days of the Last Dose of Study Drug
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 599 | 601
Participants | 12 | 17
Statistical Analysis 1: Comparison: Methylprednisolone Arm vs Placebo Arm; Test type: Superiority — It was estimated that 1200 patients (600 per trial group) would provide the trial with more than 90% power to detect superiority of methylprednisolone; p = 0.428, Regression, Logistic; Adjusted Odds Ratio = 0.74, 95% CI 2-sided [0.34 to 1.57]

3. Secondary Outcome: Number of Participants With Death or Major Complication as Defined by an Outcome in One of the 7 Highest Global Ranking Categories
Description: The 7 highest global ranking categories range from 91 (postoperative length of hospital stay > 90 days) to 97 (operative mortality).
Time Frame: Until hospital discharge, up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 599 | 601
Participants | 103 | 122
Statistical Analysis 1: Comparison: Methylprednisolone Arm vs Placebo Arm; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.228, Regression, Logistic; Adjusted Odds Ratio = 0.83, 95% CI 2-sided [0.61 to 1.13]

4. Secondary Outcome: Number of Participants With a Post-operative Length of Stay Greater Than 90 Days
Description: Calculated as discharge date minus surgery date.
Time Frame: Until hospital discharge, up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 599 | 601
Participants | 18 | 29
Statistical Analysis 1: Comparison: Methylprednisolone Arm vs Placebo Arm; Test type: Superiority — It was estimated that 1200 patients (600 per trial group) would provide the trial with more than 90% power to detect superiority of methylprednisolone over placebo; Percent Difference = -1.8, 95% CI 2-sided [-4.0 to 0.4]

5. Secondary Outcome: Number of Participants With Prolonged Mechanical Ventilation (Greater Than 7 Days)
Time Frame: Until hospital discharge, up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 599 | 601
Participants | 41 | 51
Statistical Analysis 1: Comparison: Methylprednisolone Arm vs Placebo Arm; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.309, Regression, Logistic; Adjusted Odds Ratio = 0.79, 95% CI 2-sided [0.50 to 1.25]

6. Secondary Outcome: Number of Participants With Post-operative Low Cardiac Output Syndrome
Description: Based upon the STS-CHSD registry defined "cardiac dysfunction resulting in low cardiac output" complication variable.
Time Frame: Until hospital discharge, up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 599 | 601
Participants | 31 | 37
Statistical Analysis 1: Comparison: Methylprednisolone Arm vs Placebo Arm; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.723, Regression, Logistic; Adjusted Odds Ratio = 0.91, 95% CI 2-sided [0.52 to 1.57]

7. Secondary Outcome: Number of Participants With Occurrence of Any One or More of the Following STS-CHSD-defined Major Post-operative Infectious Complications: Postprocedural Infective Endocarditis, Pneumonia, Sepsis, Deep Wound Infection, Mediastinitis.
Time Frame: Until hospital discharge, up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 599 | 601
Participants | 31 | 24

8. Secondary Outcome: Number of Participants With Any Other Post-operative Complications From the Start of Study Drug Administration Until Hospital Discharge.
Time Frame: Until hospital discharge, up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 599 | 601
Participants | 237 | 264
Statistical Analysis 1: Comparison: Methylprednisolone Arm vs Placebo Arm; Test type: Superiority; p = 0.256, Regression, Logistic; Adjusted Odds Ratio = 0.86, 95% CI 2-sided [0.67 to 1.11]

9. Secondary Outcome: PK/PD - Time to Maximum Concentration (Tmax)
Time Frame: Pre-2nd dose and minimum of 2 of any of the following 5 time points (0-30 minutes after the start of CPB, 0-30 minutes after MUF, 1-2 hours after completion of CPB, 4-6 hours after completion of CPB, or 16-24 hours after completion of CPB)
Population: Data not collected.
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: PK/PD - Maximum Concentration (Cmax)
Time Frame: as for outcome 9
Population: Data not collected.
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: PK/PD - Clearance (CL)
Time Frame: as for outcome 9
Population: Data not collected.
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: PK/PD - Volume of Distribution (Vd)
Time Frame: as for outcome 9
Population: Data not collected.
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Post-operative Biomarkers of the Inflammatory Response to Cardiopulmonary Bypass Including Interleukins 6 and 8
Description: Only to be collected at select centers and in those patients whose parent/legally authorized representative have granted consent to blood draws
Time Frame: Pre-2nd dose; a minimum of 2 of any of the following 5 time points (0-30 min after the start of CPB, 0-30 min after MUF, 1-2 hrs after CPB end, 4-6 hrs after CPB end, or 16-24 hrs after CPB end); and 36-48 hrs after CPB end
Population: Data not collected.
Arm/Group | Methylprednisolone Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Until hospital discharge, up to 4 months
Arm/Group | Methylprednisolone Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 12/599 | 17/601
Serious Adverse Events (participants affected / at risk) | 2/599 | 0/601
Other Adverse Events (participants affected / at risk) | 155/599 | 176/601
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylprednisolone Arm (N=599) | Placebo Arm (N=601)
Cardiac dysfunction (Cardiac disorders) | 1 | 0 — Study drug-related.
Hypotension (Vascular disorders) | 1 | 0 — Study drug-related.
Enterovirus infection (Infections and infestations) | 1 | 0 — Study drug-related.
Rhinovirus infection (Infections and infestations) | 1 | 0 — Study drug-related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylprednisolone Arm (N=599) | Placebo Arm (N=601)
Arrhythmia (Cardiac disorders) | 155 | 176
Cardiac dysfunction (Cardiac disorders) | 133 | 135
Cardiac Arrest (Cardiac disorders) | 31 | 37
Pericardial effusion (Cardiac disorders) | 14 | 21
Intracardiac thrombus (Cardiac disorders) | 2 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 125 | 135
Procedural complication (Injury, poisoning and procedural complications) | 41 | 42
Wound dehiscence (Injury, poisoning and procedural complications) | 11 | 9
Subdural haemorrhage (Injury, poisoning and procedural complications) | 4 | 3
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 74 | 83
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 36 | 37
Vocal cord dysfunction (Skin and subcutaneous tissue disorders) | 27 | 35
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 | 27
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 15 | 19
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Pulmonary hypertensive crisis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac operation (Surgical and medical procedures) | 30 | 35
Ventricular assist device insertion (Surgical and medical procedures) | 31 | 25
Hospitalization (Surgical and medical procedures) | 19 | 27
Cardiac pacemaker insertion (Surgical and medical procedures) | 7 | 8
Wound infection (Infections and infestations) | 14 | 21
Sepsis (Infections and infestations) | 22 | 11
Pneumonia (Infections and infestations) | 7 | 11
Mediastinitis (Infections and infestations) | 4 | 3
Venous occlusion (Vascular disorders) | 12 | 19
Haemorrhage (Vascular disorders) | 7 | 21
Deep vein thrombsis (Vascular disorders) | 7 | 14
Catheterization cardiac (Investigations) | 22 | 33
Seizure (Nervous system disorders) | 11 | 13
Cerebrovascular accident (Nervous system disorders) | 10 | 6
Nervous system disorder (Nervous system disorders) | 2 | 3
Intraventricular haemorrhage (Nervous system disorders) | 1 | 2
Multiple organ dysfunction syndrome (General disorders) | 3 | 6
Acute kidney injury (Renal and urinary disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT03229538/Prot_SAP_001.pdf
  • Informed Consent Form (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT03229538/ICF_002.pdf